CLINICAL TRIAL: NCT03904875
Title: Impact of Air Pollution on Chronic Obstructive Pulmonary Disease (COPD) Exacerbation in Haut de France. BePoPi Project.
Brief Title: Air Pollution and COPD Exacerbation
Acronym: BePoPi
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: Clinique de l'Europe, Amiens (Unknown); University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: PI2019_843_0008
Record Dates: First submitted 2019-04-04; First posted 2019-04-05 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Pollution; Exposure; Chronic Obstructive Pulmonary Disease
Keywords: pollution; Chronic Obstructive Pulmonary Disease; ultrathin particles
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: collection of data about each acute exacerbation of COPD — COPD is chronic obstructive pulmonary disease. Data collected are need of hospitalisation, final diagnosis, home address, work address and air quality data.

SUMMARY:
There is an excess of hospitalization rates for acute exacerbation of COPD in Picardy compared to the national data. A first study realized in Picardy has shown a link between air quality and COPD. Nevertheless, the particles type is unknown and according to it, impact on COPD could be different. The investigator goal is to find a correlation between acute exacerbation of COPD consultation rate and daily ultra thin particles in Haut de France. The investigators will correlate the particles composition with daily acute exacerbation of COPD rate. All COPD patients with a diagnosis of acute exacerbation in emergency room in University Hospital of Amiens-Picardie and Lille, and Clinique de l'Europe between 01/01/2020 and 31/12/2020 will be included. For each patient, home and work address will be collected. The duration of 1 year was chosen to take into account seasonal variations. In parallel, a daily report of the rate of ozone, particles (PM2.5 and PM10), dioxide nitrogen but also odours and pollens will be done by ATMO Haut de France.

ELIGIBILITY:
Inclusion Criteria:

* COPD patients with a diagnosis of acute exacerbation of COPD in the emergency room of Amiens and Lille centers
* Adults
* Patients able to express consent
* signed written informed consent form
* covered by national health insurance

Exclusion Criteria:

* patients non covered by national health insurance
* patients not able to express consent
* minors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All COPD patients with a diagnosis of acute exacerbation in emergency room in University Hospital of Amiens-Picardie and Lille, and Clinique de l'Europe between 01/01/2020 and 31/12/2020 will be included. Home and work address and spirometric data will be collected. Atmo Hauts-de-France will collect daily data on PM10, PM2,5, NO2 et O3 in Amiens and Lille metropoles. Odours and pollens will be collected too by ATMO Haut de France.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-03-12 (Actual); Study Completion 2023-09-12 (Actual)

PRIMARY OUTCOMES:
daily rate of COPD exacerbation consultation in the emergency room of the 3 centers | every day during 12 months
  daily rate of COPD exacerbation consultation in the emergency room of the 3 centers
ultrathin particles quantity in the air | every day during 12 months
  ultrathin particles quantity will be determined by the air of "Haut de France" by the company ATMO Haut de France.

SECONDARY OUTCOMES:
chemical composition ultrathin particles | every day during 12 months
  chemical composition ultrathin particles will be determined by the air of "Haut de France" by the company ATMO Haut de France.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France